CLINICAL TRIAL: NCT05918380
Title: ACHIEVE GREATER: Addressing Cardiometabolic Health In Populations Through Early Prevention in the Great Lakes Region
Brief Title: Project 3: ACHIEVE- CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Sanjay Rajagopalan, Chief, Cardiovascular Medicine, Chief Academic and Scientific Officer, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20220763
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Coronary Heart Disease
Keywords: Health Disparities; African American; Prevention; Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Motion Pictures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low CVD risk (Other): PAL2
  Interventions: Behavioral: PAL2
- High CVD risk (Other): Center for Integrated and Novel Approaches in Vascular-Metabolic Disease (CINEMA)
  Interventions: Other: CINEMA

INTERVENTIONS:
Behavioral: PAL2 — Low CVD risk participants (CAC < 100) will be followed by their primary care provider accompanied by monthly contact with community health workers provided by ACHIEVE Greater who will screen participants for social determinants of health and implement the PAL2.
  PAL2 is defined as a community health worked based intervention to mitigate psychosocial and health equity barriers to optimize health promotion coupled with high blood pressure and lifestyle disease state education.
  Other Names: Pragmatic personalized, adaptable approach to lifestyle and life circumstance
  Arms: Low CVD risk
Other: CINEMA — High CVD risk participants (CAC ≥ 100) will be followed by specialists in the Center for Integrated and Novel Approaches in Vascular-Metabolic Disease (CINEMA) at UHCMC. While they too will be assessed, by the CHW for SDOH and a plan developed to address them, this plan will be addressed by the usual resources available in the CINEMA clinic.
  Arms: High CVD risk

SUMMARY:
This project is part of the ACHIEVE GREATER (Addressing Cardiometabolic Health In Populations Through Early Prevention in the Great Lakes Region) Center (IRB 100221MP2A), the purpose of which is to reduce cardiometabolic health disparities and downstream Black-White lifespan inequality in two cities: Detroit, Michigan, and Cleveland, Ohio. The ACHIEVE GREATER Center will involve three separate but related projects that aim to mitigate health disparities in risk factor control for three chronic conditions, hypertension (HTN, Project 1), heart failure (HF, Project 2) and coronary heart disease (CHD, Project 3), which drive downstream lifespan inequality. All three projects will involve the use of Community Health Workers (CHWs) to deliver an evidence-based practice intervention program called PAL2. All three projects will also utilize the PAL2 Implementation Intervention (PAL2-II), which is a set of structured training and evaluation strategies designed to optimize CHW competence and adherence (i.e., fidelity) to the PAL2 intervention program. The present study is Project 3 of the ACHIEVE GREATER Center.

ELIGIBILITY:
Inclusion Criteria:

1. 40 to 75 years of age
2. Self-identified as Black or African American
3. Residence in the Cleveland Metro Area
4. Must have at least two of the following risk factors identified at a UH health fair screenings, with one risk factor being with SBP, A1c, or LDL:

   1. BMI≥30 mg/dL
   2. History of smoking
   3. Elevated blood pressure defined as SBP>140 or DBP>80 mmHg
   4. HbA1c≥5.7%
   5. LDL≥130
5. Able to complete a coronary artery calcium score test (CAC)
6. Willing and able to consent
7. Willing to have a UH provider and UH care
8. Currently insured for standard of care procedures

Exclusion Criteria:

1. Established documented cardiovascular disease (coronary artery disease, peripheral artery disease, myocardial infarction, stroke).
2. Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg
3. Lung disease requiring supplemental oxygen therapy
4. Individuals receiving treatment for cancer related disease
5. Pregnant or nursing mothers

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Triple Goal | 12 months
  Percent reaching triple goal of BP <130/80 mm Hg, HbA1c<5.7% and LDL-C <130 mg/dl (<100 if high-risk)

SECONDARY OUTCOMES:
Change in HbA1c as measured by blood work | baseline, 12 months
  Percent change in HbA1c
Change in LDL-C as measured by blood work | baseline, 12 months
  Percent change in LDL-C
Change in blood pressure | baseline, 12 months
  Percent change in blood pressure
Change in weight | baseline, 12 months
  Percent change in weight

OTHER OUTCOMES:
Health Visits and Lifestyle Changes - Medical/Mental Health Visits | 12 months after cessation of intervention or 24 months after enrollment
  1-year rate of new medical/mental health visits
Health Visits and Lifestyle Changes - Smoking Cessation | 12 months after cessation of intervention or 24 months after enrollment
  1-year rate of smoking cessation
Health Visits and Lifestyle Changes - Diet | 12 months after cessation of intervention or 24 months after enrollment
  1-year rate of changes in diet
Health Visits and Lifestyle Changes - Activity | 12 months after cessation of intervention or 24 months after enrollment
  1-year rate of changes in activity

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajagopalan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No